CLINICAL TRIAL: NCT03153254
Title: Usability Study of an Active Smart Wearable Orthosis for Enhanched Rehabilitation Therapy in Stroke Patients
Brief Title: Active Smart Wearable Orthosis for Enhanched Rehabilitation THErapy
Acronym: ARTHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas More Kempen (Other)
Collaborators: Ortho-Medico (Unknown)
Responsible Party: Principal Investigator, Lieven De Maesschalck, Innovation Manager, Thomas More Kempen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: S60144
Record Dates: First submitted 2017-03-06; First posted 2017-05-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: Upper extremity; Rehabilitation; Robot assisted therapy; Robotics; Devices; Orthosis
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: Phase 1: Healthy persons Phase 2: Stroke patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy persons (Experimental): Test upper limb robot assisted therapy device. During 1 session of 1/2 hour.
  Interventions: Device: Test upper limb robot assisted therapy device
- Stroke patients (Experimental): Training with new upper limb robot assisted therapy device. During 2 to 5 sessions of 1/2 hour.
  Interventions: Device: Training with new upper limb robot assisted therapy device

INTERVENTIONS:
Device: Test upper limb robot assisted therapy device — During 1 session of 1/2 hour.
  Other Names: active orthosis; exoskeleton
  Arms: Healthy persons
Device: Training with new upper limb robot assisted therapy device — During 2 to 5 sessions of 1/2 hour.
  Other Names: active orthosis; exoskeleton
  Arms: Stroke patients

SUMMARY:
The purpose of this study is to investigate the usability of a new upper limb robot assisted therapy device in stroke patients.

DETAILED DESCRIPTION:
The number of physically weak individuals is increasing, resulting in a higher burden on health care and health care workers. The use of robot assisted therapy (RAT) might partly solve this problem. Rehabilitation progress highly depends on training intensity and training duration, favouring the use of RAT.

In this pilot study, the usability of a new upper arm RAT device for upper arm rehabilitation in stroke patients is investigated. Myo-electrical signals will serve as input for the device, assisting the user in flexion and extension of the elbow, which is combined with a stabilizing shoulder brace and a bionic glove.

ELIGIBILITY:
1. Healthy subjects:

   Inclusion criteria:
   * Persons between 18 and 85 years old that can perform all sorts of daily activities with their upper limbs
   * Ability to sit on a chair with adequate trunk stability
   * Ability to follow verbal instructions
   * Ability to communicate verbally with the researchers

   Exclusion criteria:
   * Ever had a fracture in the upper limbs
   * Ever had a surgery in the upper limbs
   * Pain in the upper limbs obstructing the execution of daily activities with the upper limbs
   * Physical trauma in the two months preceding the research
   * Mental problems that make the execution of daily activities unreliable
   * (Chronic) subluxation of the shoulder joint
   * Secundary soft tissue problems which may complicate the research or make it impossible (e.g. shoulder impingement, musculoskeletal problems, sensory deficits)
   * Pregnancy
   * Pacemaker
   * Known allergies for one of the components of the ARTHE rehabilitation tool
2. Stroke patients:

Inclusion criteria:

* Stroke patients, more than three months after onset
* Aged between 18 and 85 years
* None to moderate spasticity in the hemiplegic arm (Modified Ashworth Scale: 0-2)
* Detectable voluntary muscle activity at elbow flexion and elbow extension of the hemiplegic arm (Medical research council score: 1-5)
* Ability to sit on a chair with adequate trunk stability
* Ability to follow verbal instructions
* Ability to communicate verbally with the researchers

Exclusion criteria:

* Stroke patients, less than three months after onset
* Massive spastic patterns
* Severe medical conditions that interfere with the proper execution of the research, patients who are medically unstable
* Cognitive disorders which may complicate the research or make it impossible
* Speaking disorders (aphasia, dysarthria) which may complicate the proper execution of the research and the communication of important verbal information
* Visual disorders which may complicate the research or make it impossible
* (Chronic) subluxation of the shoulder joint
* Shoulder-hand-syndrom
* Pusher syndrom
* Secundary soft tissue problems which may complicate the research or make it impossible (e.g. shoulder impingement, musculoskeletal problems, sensory deficits)
* Pregnancy
* Pacemaker
* Known allergies for one of the components of the ARTHE rehabilitation tool

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Investigate user experience by a self-composed questionnaire. | Up to 30 minutes at the last session
  Investigate user experience by a self-composed questionnaire with theorems where upon users have to score. Possible scores range from 1 (totally disagree) to 4 (totally agree).

SECONDARY OUTCOMES:
Measure the rate of perceived exertion by the Borg scale. | Up to 5 minutes at the last session
  Measure the rate of perceived exertion by the Borg scale. The Borg scale is a way of measuring physical activity intensity level. Possible scores range from 0 (no fatigue at all) to 10 (worst imaginable fatigue).
Investigate whether wearing the device improves functionality by the Action Research Arm Test (ARAT). | Up to 5 weeks (at week 1, week 2 and week 5)
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven De Maesschalck, Principal Investigator — Thomas More Kempen
Locations (4):
- Belgium (4):
  - RevArthe, Edegem, Antwerp
  - Thomas More - Mobilab, Geel, Antwerp
  - REVAlution, Herentals, Antwerp
  - Revalidatie & MS Centrum, Overpelt, Antwerp

IPD SHARING:
Plan to Share IPD: No